CLINICAL TRIAL: NCT03341897
Title: Endovasculer Treatement of Male Pelvic Venous Insufficiency
Brief Title: Varicocele Treatement by Endovasculer Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VARICOCELE TREATEMENT
Record Dates: First submitted 2017-10-03; First posted 2017-11-14 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Varicocele
Keywords: embolization; coiling; varicocele
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical varicocelectomy (Experimental)
  Interventions: Procedure: endovasculer embolization of varicocele

INTERVENTIONS:
Procedure: endovasculer embolization of varicocele — Step 1: Vascular Access
  Access can be achieved via the internal jugular or femoral veins. Step 2: Left Renal Vein Injection Step 3: Left Spermatic Vein Catheterization Step 4: Spermatic Vein Occlusion Step 5: Right Spermatic Venography POSTPROCEDURE CARE
  The patient is kept in bed for 1 hour postprocedure. The patient is advised to take anti-inflammatory agents as needed and to avoid any activity involving the Valsalva maneuver, such as lifting, vigorous, or "hitting type" sports for 3 full days beginning the day after the proce¬dure. Most patients report a minor dull ache in the back or groin lasting < 2 to 5 days. Fewer than 5% of patients will develop more severe pain lasting up to 14 days, requiring oral analgesics and anti-inflammatory agents and avoidance of vigorous exercise.

SUMMARY:
A varicocele is a collection of varicose veins within the pampiniform (spermatic) plexus secondary to reflux in the internal spermatic vein (ISV).The condition affects 10% to 15% of the general population but is detected in as many as 40% of men undergoing an infertility workup. Depending on the method used for diagnosis, varicoceles are reported as bilateral in 17% to 77% of men. Traditionally, the diagnosis was made through clinical examination; however,as with other venous reflux disorders, ultrasound has become the mainstay of diagnosis. The traditional indications for treatment include infertility in patients with appropriate semen abnormalities, chronic groin pain, testicular atrophy in adolescent varicoceles, and recurrent varicocele after previous repair. Other indications more recently described with variable strength of evidence include low serum testosterone (with or without erectile dysfunction), benign prostatic hypertrophy,enhancement of assisted fertility techniques, and recurrent first trimester pregnancy loss.Infertility affects 10% to 15% of men of reproductive age. In approximately 50%, a cause is not found. The proof that varicocele repair improves fertility remains elusive; however, there is general acceptance that treatment does improve abnormalities of semen production.The traditional measures to assess semen production are sperm motility,morphology, and total sperm count. However, sperm counts greatly vary from day to day in any individual patient, and these measures correlate poorly with infertility outcomes.

The investigators do this study to evaluate the effectiveness of endovascular therapy using coils and other sclerosing agents and compare their results with other traditonal surgical methods in treatement of varicocele.

DETAILED DESCRIPTION:
All included patients will undergo the following:

* History & examination
* Semen analysis preintervention.
* Scrotal duplex scan of testicular vessels and testicular size .

Technique:

* All interventions will be performed in the endovascular OR with set on C-ARM.
* Patient's position and comfort are issues that are important initially.

STEPS FOR SPERMATIC VENOGRAPHY AND VARICOCELE EMBOLIZATION

Step 1: Vascular Access

Access can be achieved via the internal jugular or femo¬ral veins. Our preferred method is to puncture the right internal jugular vein under ultrasound guidance.

Step 2: Left Renal Vein Injection

During left renal vein injection, the origin of the left spermatic vein is noted .

Step 3: Left Spermatic Vein Catheterization

The catheter is manipulated into the left spermatic vein. A varicocele is present if the contrast refluxes into the pampiniform plexus. If the direction of flow is antegrade, this is considered to represent a negative spermatic venogram.

Step 4: Spermatic Vein Occlusion

If varicocele is confirmed, the spermatic vein is occluded, preferably immediately above the internal inguinal ring and along its full length to within 2 to 3 cm of its origin. The use of liquid embolics with or without metallic coils has become the most common method. Embolization with coils alone without liquid should be avoided, even for "straightforward" cases due to a high rate of recurrence. It is important to look for collaterals throughout the procedure, which may only become visible after distal occlusion . These collaterals are the usual cause of technical failure or recurrence and therefore must be occluded. Options for occlusion methods are described as follows.

Some practitioners place coils in the distal ISV before injecting glue. Coils in the proximal ISV are not necessary. Avoiding injection of glue into the scrotum is essential, either by previously placed distal coils or external compression. Overinjection of glue will result in extension into the renal vein or embolization into the pulmonary artery.

Step 5: Right Spermatic Venography

The same steps performed for the left spermatic vein are repeated for the right spermatic vein, except that the right spermatic vein usually arises directly from the infe¬rior vena cava. If reflux is demonstrated, embolization is performed in the same manner as on the left. The right spermatic vein arises from the inferior vena cava at an acute angle, which can make catheterization from the femoral route especially difficult.

POSTPROCEDURE CARE

The patient is kept in bed for 1 hour postprocedure. The patient is advised to take anti-inflammatory agents as needed and to avoid any activity involving the Valsalva maneuver, such as lifting, vigorous, or "hitting type" sports for 3 full days beginning the day after the proce¬dure. Most patients report a minor dull ache in the back or groin lasting < 2 to 5 days. Fewer than 5% of patients will develop more severe pain lasting up to 14 days, requiring oral analgesics and anti-inflammatory agents and avoidance of vigorous exercise

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 40 years.
2. Grade three reflux by duplex ultrasound..
3. Recurrent varicocele after surgical treatement.

Exclusion Criteria:

* Any contraindication for endovascular therapy regarding radiation or dye or sclerosing agents.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
semen analyis criteria | 3 month
  sperm number in milion/ml
semen analysis criteria | 3 month
  sperm motility